CLINICAL TRIAL: NCT01422187
Title: A Multicenter Extension Study of Taliglucerase Alfa in Adult Subjects With Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-06-007
Expanded Access: NCT00962260 (No longer available)
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Gaucher Disease
Keywords: enzyme replacement therapy
MeSH Terms: conditions — Gaucher Disease | interventions — taliglucerase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taliglucerase alfa 30 units/kg (Experimental): Subjects randomized to receive 30 units/kg
  Interventions: Drug: Taliglucerase alfa
- Taliglucerase alfa 60 units/kg (Experimental): Subjects randomized to 60 units/kg
  Interventions: Drug: Taliglucerase alfa

INTERVENTIONS:
Drug: Taliglucerase alfa — Taliglucerase infusion every two weeks for 21 months

SUMMARY:
This is a multi-center trial to further extend the assessment of the safety and efficacy of taliglucerase alfa in adult subjects (≥18 years old) with Gaucher disease who have enrolled in Protocol PB-06-003. Subjects will continue to receive an intravenous (IV) infusion of taliglucerase alfa every two weeks. The duration of treatment will be a maximum of 21 months or until taliglucerase alfa is commercially available to the subject at the discretion of the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed Protocol PB-06-001 and enrolled in Protocol PB-06-003
* The subject signs an informed consent

Exclusion Criteria:

* Currently taking another investigational drug for any condition.
* Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the subject's compliance with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

REFERENCES:
- [Derived] Zimran A, Duran G, Giraldo P, Rosenbaum H, Giona F, Petakov M, Terreros Munoz E, Solorio-Meza SE, Cooper PA, Varughese S, Alon S, Chertkoff R. Long-term efficacy and safety results of taliglucerase alfa through 5years in adult treatment-naive patients with Gaucher disease. Blood Cells Mol Dis. 2019 Sep;78:14-21. doi: 10.1016/j.bcmd.2016.07.002. Epub 2016 Jul 18. PMID 27499018

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Adjusted: Subjects randomized to 30 units/kg but with dose increased
  Taliglucerase alfa: Taliglucerase infusion every two weeks for 21 months
Period: Overall Study
Arm/Group | Taliglucerase Alfa 30 Units/kg | Taliglucerase Alfa 60 Units/kg | Dose Adjusted
Started | 8 | 9 | 2
Completed | 7 | 8 | 2
Not Completed | 1 | 1 | 0
Not completed — Personal reason | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Taliglucerase Alfa 30 Units/kg | Taliglucerase Alfa 60 Units/kg | Dose Adjusted | Total
Number analyzed (Participants) | 8 | 9 | 2 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (13.4) | 39.9 (12.0) | 38.5 (0.7) | 41.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 8
  Male | 4 | 6 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 9 | 2 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 2 | 2 | 0 | 4
  South Africa | 0 | 0 | 1 | 1
  Italy | 0 | 1 | 0 | 1
  Serbia | 2 | 2 | 0 | 4
  Mexico | 3 | 2 | 0 | 5
  Chile | 0 | 1 | 1 | 2
  Spain | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Spleen Volume
Description: Spleen volume measured by MRI
Time Frame: 60 months
Measure: Mean (Standard Error); unit: Milliliters
Arm/Group | Taliglucerase Alfa 30 Units/kg | Taliglucerase Alfa 60 Units/kg | Dose Adjusted
Number analyzed (Participants) | 8 | 9 | 2
Milliliters
  Baseline | 2032.0 (454.9) | 1960.0 (451.7) | 2321.7 (679.6)
  Month 12 | 1522.6 (429.6) | 1063.7 (280.7) | 1677.9 (609.3)
  Month 24 | 1193.0 (320.2) | 744.9 (130.6) | 1536.3 (506.7)
  Month 36 | 1068.7 (264.6) | 634.0 (71.0) | 1256.6 (385.0)
  Month 48 | 1137.4 (314.6) | 526.8 (48.5) | 1070.0 (280.6)
  Month 60 | 1019.2 (285.3) | 516.1 (54.5) | 919.9 (180.9)

2. Secondary Outcome: Liver Volume
Description: Liver volume by MRI
Time Frame: 60 months
Measure: Mean (Standard Error); unit: Milliliters
Arm/Group | Taliglucerase Alfa 30 Units/kg | Taliglucerase Alfa 60 Units/kg | Dose Adjusted
Number analyzed (Participants) | 8 | 9 | 2
Milliliters
  Baseline | 3103.4 (324.7) | 2536.1 (170.0) | 2488.6 (206.2)
  Month 12 | 2619.3 (266.4) | 2155.2 (104.8) | 2048.0 (87.8)
  Month 24 | 2367.9 (212.8) | 1939.5 (101.5) | 2064.0 (202.5)
  Month 36 | 2429.6 (229.6) | 2010.6 (143.5) | 1959.0 (140.5)
  Month 48 | 2429.1 (283.2) | 1971.2 (179.3) | 1792.2 (143.6)
  Month 60 | 2290.9 (233.6) | 2067.7 (188.9) | 1820.8 (196.5)

3. Secondary Outcome: Platelet Count
Description: Platelet count measure annually
Time Frame: 60 months
Measure: Mean (Standard Error); unit: platelets/mm^3
Arm/Group | Taliglucerase Alfa 30 Units/kg | Taliglucerase Alfa 60 Units/kg | Dose Adjusted
Number analyzed (Participants) | 8 | 9 | 2
platelets/mm^3
  Baseline | 70975 (8700.6) | 70067 (7695.5) | 69500 (42500)
  Month 12 | 86613 (11894) | 137556 (18358) | 88000 (65000)
  Month 24 | 103250 (17008) | 168778 (23717) | 101000 (68000)
  Month 36 | 106775 (13517) | 155667 (16060) | 94500 (64500)
  Month 48 | 100643 (15314) | 184000 (16688) | 103000 (53000)
  Month 60 | 104986 (18961) | 180625 (17062) | 103500 (60500)

4. Secondary Outcome: Hemoglobin
Description: Hemoglobin measure yearly
Time Frame: 60 months
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Taliglucerase Alfa 30 Units/kg | Taliglucerase Alfa 60 Units/kg | Dose Adjusted
Number analyzed (Participants) | 8 | 9 | 2
mg/dL
  Baseline | 12.3 (0.7) | 11.6 (0.9) | 12.5 (0.9)
  Month 12 | 13.9 (0.7) | 14.2 (0.7) | 14.3 (0.9)
  Month 24 | 13.5 (0.8) | 14.1 (0.7) | 14.2 (0.2)
  Month 36 | 14.0 (0.5) | 14.2 (0.8) | 14.4 (0.1)
  Month 48 | 13.7 (0.6) | 14.0 (0.8) | 14.5 (0.1)
  Month 60 | 14.1 (0.9) | 13.9 (0.6) | 14.3 (0.1)

ADVERSE EVENTS:
Time Frame: 21 Months
Arm/Group | Taliglucerase Alfa 30 Units/kg | Taliglucerase Alfa 60 Units/kg | Dose Adjusted
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/9 | 0/2
Other Adverse Events (participants affected / at risk) | 6/8 | 8/9 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taliglucerase Alfa 30 Units/kg (N=8) | Taliglucerase Alfa 60 Units/kg (N=9) | Dose Adjusted (N=2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — right hip arthrosis which required artificial hip implantation
Thyroid Carcinoma (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — papillary thyroid carcinoma that required total thyroidectomy and left node resection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taliglucerase Alfa 30 Units/kg (N=8) | Taliglucerase Alfa 60 Units/kg (N=9) | Dose Adjusted (N=2)
NASOPHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No